CLINICAL TRIAL: NCT05420272
Title: Trunk Endurance and Performance in Pes Planus
Brief Title: Comparison of Lower Extremity Biomechanics,Core Endurance, and Performance in Pes Planus : A Controlled Study
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Tezel Yıldırım Şahan, Clinical Researcher, Hacettepe University
Other Study IDs: 2022-170
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Pes Planus
Keywords: pes planus; trunk; subtalar angle; endurance; kinect
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pes planus: Evaluation group- Trunk performance and endurance lower extremity biomechanics
  Interventions: Behavioral: Trunk performance and endurance lower extremity biomechanic
- Control group healthy: Trunk performance and endurance lower extremity biomechanics
  Interventions: Behavioral: Trunk performance and endurance lower extremity biomechanic

INTERVENTIONS:
Behavioral: Trunk performance and endurance lower extremity biomechanic — Trunk performance and endurance lower extremity biomechanic
  Other Names: asymtopamtic healthy control Trunk performance and endurance lower extremity biomechanic

SUMMARY:
Pes planus is a deformity called "flatfoot" and is defined as the valgus of the hindfoot while loading the foot, the disappearance of the medial longitudinal arch in the midfoot, and the supination of the forefoot relative to the hindfoot. The aim of this study is to compare the subtalar angle, q angle, trunk muscle endurance, and performance of individuals with pes planus and healthy controls. Volunteer students between the ages of 18-35 will be included among the students studying at the Health Sciences University Gülhane Faculty of Physiotherapy and Rehabilitation. The feet of individuals who want to be included in the study will be examined by the researchers with the navicular drop test and the presence of pes planus will be determined according to this test. Subtalar Angle to determine the degree of rotation (Varus/Valgus) in the hindfoot, Q Angle for knee biomechanics, Navicular Drop Test to determine flat feet, Mcgill trunk Flexion, Extension, and Lateral Bridge Test to evaluate trunk endurance, Xbox to evaluate lower and upper extremity performance 360Kinect™ game console will be used. In this study, statistical analyzes will be made with SPSS 21 package program (IBM Corp., Armonk, NY, USA). Wilcoxon test or Mann Whitney U will be used after determining the conformity to the normal distribution in the comparison of the values before and after the exercises, individuals with and without flat feet. Results will be evaluated at the significance level of p<0.05. Cohen's d values will be calculated to determine the study effect size.

DETAILED DESCRIPTION:
The navicular drop test is a test used to measure the amount of pronation in the foot, which is obtained by subtracting the navicular height measured while standing with weight on the foot, from the navicular height measured in the sitting position without placing weight on the foot. While individuals are sitting on a chair with bare feet, the navicular tubercle will be marked on both feet and marked at the level of the navicular tubercle on a card on the floor. Then, the individual will be asked to stand up, and the navicular tubercle level will be marked again on the same card while giving full weight to the foot. The expression in millimeters of the distance between both lines will be recorded as the amount of navicular drop. The amount of navicular drop between 6 and 9 millimeters will be considered as normal MLA, and if it is 10 millimeters or more, it will be considered as pes planus. This test will be done for both the right foot and the left foot To measure the subtalar angle, the participants will be asked to lie face down with their feet hanging out of the bed. The subtalar neutral position (without the foot in pronation or supination) will be determined, and the calcaneal midline and the distal 1/3 tibial longitudinal midline will be marked with a line. The pivot point of the goniometer will be placed on the midline of the Achilles tendon and one arm will reference the distal 1/3 tibial longitudinal midline while one arm will refer to the calcaneal line and the deviation angle will be recorded. The deviation angle in the valgus direction will be given a negative (-) value, and the deviation angle in the varus direction will be given a positive (+) value. This measurement will be made for both the right foot and the left foot The Q angle is the angle between the line extending from the anterior superior iliac spine to the middle of the patella and the line drawn from the middle of the patella to the tibial tubercle. Measurements will be made by means of a goniometer. Its normal value is 8-14° (average 10°) in men and 11-20° (mean 15°) in women. Right Q angle and left Q angle will be measured with the patient in the supine position and without contracting the quadriceps Mcgill trunk flexion test is a test used to evaluate the endurance of trunk flexor muscles, McGill trunk extension test trunk extensor muscles, McGill lateral bridge test is a test used to evaluate the endurance of core muscles that provide lateral stability. In the Mcgill trunk flexion test, participants will be asked to cross their hands on their chest and will be positioned on the floor with their trunks flexed at 60° and their knees flexed at 90°. Sixty degrees of body flexion will be provided by a stretcher with an adjustable head. It will be ensured that there is no support behind the person during the test. In the Mcgill trunk extension test, the participants will be positioned in the prone position with their spina iliaca anterior superior to the side of the bed. Participants will be asked to extend their upper body straight forward from the edge of the table and will be fixed above their knees with the help of a belt. Before the test starts, the upper extremity will be supported with the help of a stool placed on the floor to prevent fatigue. When ready for the test, the participant will be asked to raise their hands on the stool and cross them in front of their torso and stand parallel to the ground. In the Mcgill lateral bridge test, the participants will lie on their dominant side, place their foot on the other foot, cross their non-dominant arm over their chest and place them on the dominant shoulder, and the dominant forearm shoulder straps. The participant will be asked to stand on the elbow. As soon as the participant is ready, he will be asked to stand on his forearm with his body on a single line, and the stopwatch will be started, which will raise his hips. The person will be asked to maintain the positions for as long as possible. Before the tests, individuals will be shown how to do the tests and they will be given a trial for a few seconds. The stopwatch will be started and the test will be started, in case of any deterioration in its position, the stopwatch will be stopped and the test will be terminated. The elapsed time will be recorded in seconds. Mcgill trunk flexion-extension and lateral bridge tests were previously performed in healthy individuals and their validity and reliability were found to be high. (McGill trunk flexion intra-class correlation coefficient (ICC) = 0.97, McGill trunk extension intra-class correlation coefficient (ICC) = 0.97, McGill lateral bridge intra-class correlation coefficient (ICC) = 0.99) (37.38.39).

Xbox 360Kinect™ game console was used for upper and lower extremity performance evaluation. Xbox Kinect; There is an infrared Kinect camera sensor that can detect user movements without the need for a special controller, the movements of the user in the virtual reality environment can be monitored in real-time on the screen. Before starting the play therapy, the patients were informed about the games by the physiotherapist and they were shown how to play the games. 100 m running game in Kinect Sport for 100 m running performance, single-leg jump game in Kinect Sport for single-leg jump performance, discus throw game for upper extremity performance. will be determined and the scores of the participants will be recorded. Kinect is a valid and reliable method for evaluating upper and lower extremity function In this study, statistical analyzes will be made with SPSS 21 package program (IBM Corp., Armonk, NY, USA). Wilcoxon test or Mann Whitney U will be used after determining the conformity to the normal distribution in the comparison of the values before and after the exercises, individuals with and without flat feet. Results will be evaluated at the significance level of p<0.05. Cohen's d values will be calculated to determine the study effect size.

ELIGIBILITY:
Inclusion Criteria:

* Being 18-35 years
* Being a volunteer to participate in the study.

Exclusion Criteria:

* Individuals who have had any previous surgery related to the lower extremities, who have any orthopedic, neurological, and systemic problems that may affect the lower extremity and balance, and those with congenital shortness of the lower extremities and visual impairment will be excluded from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pes planus
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Comparison of Trunk endurance in pes planus and controls | 10 minute
  Trunk endurance

SECONDARY OUTCOMES:
Comparison of Subtalar Angle, q angle | 10 minute
  subtalar angle , q angle
comparison of trunk performance | 10 minute
  kinect performance test

CONTACTS AND LOCATIONS:
Overall Officials: Tezel Y Şahan, pHD, Study Chair — University of Health science
Locations (1):
- University of Health Science, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The authors can want from the corresponding author from journals system.

REFERENCES:
- [Background] Gün, K., M. SaridoĞan, and Ö. Uysal, Pes Planus Tanısında Ayak İzi ve Radyografik Ölçüm Yöntemlerinin Korelasyonu. Turkish Journal of Physical Medicine & Rehabilitation/Turkiye Fiziksel Tip ve Rehabilitasyon Dergisi, 2012. 58(4).
- [Background] Milenković, S., et al., Incidence of flat foot in high school students. Facta universitatis-series: Physical Education and Sport, 2011. 9(3): p. 275-281.
- [Background] Aenumulapalli A, Kulkarni MM, Gandotra AR. Prevalence of Flexible Flat Foot in Adults: A Cross-sectional Study. J Clin Diagn Res. 2017 Jun;11(6):AC17-AC20. doi: 10.7860/JCDR/2017/26566.10059. Epub 2017 Jun 1. PMID 28764143
- [Background] Shih YF, Chen CY, Chen WY, Lin HC. Lower extremity kinematics in children with and without flexible flatfoot: a comparative study. BMC Musculoskelet Disord. 2012 Mar 2;13:31. doi: 10.1186/1471-2474-13-31. PMID 22381254